CLINICAL TRIAL: NCT04887727
Title: Development of Oral Amino Acid Tracers to Study Protein Turnover in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Daniel Moore, Associate Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Connaught
Record Dates: First submitted 2021-05-05; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Healthy Adult Males

STUDY DESIGN:
Intervention Model Description: Three groups: Fast, Fed, Ex-Fed Two trials per group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy, recreationally-active adult males - Muscle Trial (Experimental): Subjects receive 0.25g/kg crystalline amino acids modelled after egg protein, enriched with L-[1-13C]leucine and L-ring-[2H5]phenylalanine with a primed-constant infusion of L-[555-2H3]leucine to assess myofibrillar protein synthesis rates
  Interventions: Dietary Supplement: Crystalline amino acids to assess myofibrillar protein synthesis rates
- Healthy, recreationally-active adult males - Whole Body Trial (Experimental): Subjects receive 0.25g/kg crystalline amino acids modelled after egg protein, enriched with L-[1-13C]leucine with a primed-constant infusion of L-[555-2H3]leucine to whole-body protein turnover, amino acid oxidation, and net protein balance
  Interventions: Dietary Supplement: Crystalline amino acids to assess whole-body protein turnover, amino acid oxidation, and net protein balance

INTERVENTIONS:
Dietary Supplement: Crystalline amino acids to assess myofibrillar protein synthesis rates — Amino acid dose = 0.25g/kg bodyweight
  Arms: Healthy, recreationally-active adult males - Muscle Trial
Dietary Supplement: Crystalline amino acids to assess whole-body protein turnover, amino acid oxidation, and net protein balance — Amino acid dose = 0.25g/kg bodyweight
  Arms: Healthy, recreationally-active adult males - Whole Body Trial

SUMMARY:
Previous studies have used a combination of oral L-[1-13C]leucine and intravenous labeled L-[5,5,5-2H3]leucine to assess the acute postprandial changes in whole-body protein turnover (12, 19). Intravenous and dietary-labeled amino acid tracers have also been used in tandem to assess rates of myofibrillar protein synthesis in response to bolus protein ingestion and resistance exercise (46). By validating whole-body net balance to myofibrillar protein synthesis, our proposed multi-tracer approach will develop minimally invasive models to study protein turnover in a variety of populations in which traditional infusions and/or repeated blood samples are not possible (i.e. pediatric, free-living populations).

DETAILED DESCRIPTION:
The primary objective of the proposed study is to validate the use of a novel oral tracer model to accurately and reliably measure myofibrillar protein synthesis. It is hypothesized that oral L-[1-13C]leucine and L-[ring-2H5]phenylalanine, ingested as a bolus to mimic an intravenous 'pulse dose' administration (51, 65), will reveal similar rates of myofibrillar protein synthesis when compared to traditional intravenous L-[5,5,5-2H3]leucine infusion. Moreover, it is hypothesized that both methods will reveal the expected graded changes in myofibrillar protein synthesis in response to feeding and resistance exercise (i.e. fasted<feeding<exercise & feeding).

The secondary objective of the proposed study is to develop and validate non-invasive models to measure whole-body amino acid oxidation and net balance in response to feeding and resistance exercise. It is hypothesized that whole-body net balance, as determined by a novel oral tracer model (i.e. L-[1-13C]leucine) , will align with traditional intravenous tracer methodology (i.e. L-[5,5,5-2H3]leucine) and reveal the expected physiological changes in whole-body protein turnover in response to feeding and resistance exercise (i.e. fasted<feeding<exercise & feeding).

ELIGIBILITY:
Inclusion Criteria:

* Male
* Currently performing structured physical activity 2-5 days per week

Exclusion Criteria:

* Unable to safely perform exercise as per PARQ+ guidelines
* Currently using tobacco products
* Currently using or have history of anabolic steroid use
* Diagnosed with medical condition including type 2 diabetes, cancer, heart disease
* Unable to abstain from supplement use (HMB, branched chain amino acids, phosphatidic acid) for at least three weeks prior to trial
* currently using medications known to affect protein metabolism e.g. corticosteroids, NSAID, prescription-strength acne medication
* allergic to local anesthetics
* female: Hormonal fluctuations associated with the menstrual cycle have been reported to alter protein metabolism during exercise and may influence indices of the post-exercise myofibrillar protein synthetic response. Accordingly, the study will include males to ensure a stable hormonal environment and to increase the homogeneity of the physiological response.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Myofibrillar protein synthesis rates | 5 hours
  Myofibrillar protein synthesis rates assessed by oral and intravenous tracers during Fast, Fed, and Ex-Fed

SECONDARY OUTCOMES:
Whole-body protein turnover | 5 hours
  Whole-body protein turnover assessed by oral and intravenous tracers during Fast, Fed, and Ex-Fed
Amino acid oxidation and net protein balance | 5 hours
  Amino acid oxidation and net protein balance assessed by oral tracers during Fast, Fed, and Ex-Fed. Net protein balance is derived from the difference between amino acid intake (known) and total amino acid oxidation over the 5h measurement period.
Muscle anabolic signalling | 2 and 5 hours
  Immunoblotting for mTORC1/key downstream targets of mTORC1
Amino acid transporter expression | 2 and 5 hours
  Immunoblotting for amino acid transporters LAT1/SNAT2

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Moore, PhD, Principal Investigator — University of Toronto
Locations (1):
- Goldring Centre for High Performance Sport at the University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mazzulla M, Hodson N, West DWD, Kumbhare DA, Moore DR. A non-invasive 13CO2 breath test detects differences in anabolic sensitivity with feeding and heavy resistance exercise in healthy young males: a randomized control trial. Appl Physiol Nutr Metab. 2022 Aug 1;47(8):860-870. doi: 10.1139/apnm-2021-0808. Epub 2022 May 24. PMID 35609328